CLINICAL TRIAL: NCT04314037
Title: A Phase I, Open-label, Randomized, Four-period, Crossover, Fully Replicated, Reference-scaled, Single Center Study to Assess the Bioequivalence of a Single Oral Dose of 1200 mg of the Coated Cesol Tablet Formulation Versus Comparator Biltricide® in Healthy Male Volunteers
Brief Title: Bioequivalence Study of Coated Cesol Tablet Formulation Versus Biltricide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200585_0004; 2019-002868-27 (EudraCT Number)
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Bioavailability; Bioequivalence; Praziquantel; Cesol; Pharmacokinetics
MeSH Terms: interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (T1-R1-T2-R2) (Experimental): Participants will receive first dose of Cesol on Day 1 in treatment period 1 followed by first dose of Biltricide on Day 8 in treatment period 2 followed by second dose of Cesol on Day 15 in treatment period 3 followed by second dose of Biltricide on Day 22 in treatment period 4. A washout period of 7 days will be maintained between 4 treatment periods.
  Interventions: Drug: Cesol (Test); Drug: Biltricide (Reference)
- Sequence 2 (R1-T1-R2-T2) (Experimental): Participants will receive first dose of Biltricide on Day 1 in treatment period 1 followed by first dose of Cesol on Day 8 in treatment period 2 followed by second dose of Biltricide on Day 15 in treatment period 3 followed by second dose of Cesol on Day 22 in treatment period 4. A washout period of 7 days will be maintained between 4 treatment periods.
  Interventions: Drug: Cesol (Test); Drug: Biltricide (Reference)

INTERVENTIONS:
Drug: Cesol (Test) — Participant will receive coated cesol tablet in sequence 1 (Day 1 and Day 15) and in sequence 2 (Day 8 and Day 22). A washout period of 7 days will be maintained between 4 treatment periods.
  Other Names: Praziquantel
Drug: Biltricide (Reference) — Participant will receive biltricide tablet in Sequence 1 (Day 8 and Day 22) and in sequence 2 (Day 1 and Day 15). A washout period of 7 days will be maintained between 4 treatment periods.
  Other Names: Praziquantel

SUMMARY:
The purpose of this study is to assess the bioequivalence (BE) of new coated Cesol tablet (Test) versus Biltricide tablets (Comparator) in healthy male participants. Praziquantel (rac-PZQ) is the active ingredient for Cesol and Biltricide tablets.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring
* Nonsmoker (=0 cigarettes, pipes, cigars or others) since at least 3 months
* Have a body weight within 55.0 to 95.0 kilogram (kg) and body mass index within the range of 18.5 to 29.9 kilogram per meter squared (kg/m^2)
* Electrocardiogram recording (12-lead) without signs of clinically relevant pathology in particular heart-rate corrected [QTc] (Bazett) <450 milliseconds (ms)
* Vital signs should be in normal range (systolic blood pressure: 90 to 140 millimeters of mercury [mmHg]; diastolic blood pressure: 50 to 90 mmHg; pulse rate: 50 to 90 beats per minute [bpm]; auricular body temperature between 35.9 degree centigrade [°C] to 37.6°C)
* Are males agreeing to refrain from donating sperm, Use a male condom when having sexual intercourse with a woman of child-bearing potential, who is not currently pregnant, and advise her to use a highly effective contraceptive method with a failure rate of less than (< )1 percent (%) per year
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Any condition, including any clinically relevant abnormality in the safety laboratory parameters as judged by the Investigator, that in the Investigator's opinion constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
* Have positive results from serology examination for Hepatitis B surface antigen (indicative of active Hepatitis B), Hepatitis C Virus or Human Immunodeficiency Virus (Human Immunodeficiency Virus 1/2 antibodies)
* Participants who have used drugs that may affect the pharmacokinetics of rac-PZQ from 15 days before dosing until the last PK sample, example., phenytoin, barbiturates, primidone, carbamazapine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, oral ketoconazole
* Positive test for drugs of abuse (including alcohol) at Screening and prior to each dosing
* Unlikely to comply with the protocol requirements, instructions and study-related restrictions; example, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study
* Participant is the Principal Investigator or any Sub investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study
* Inability to communicate or cooperate with the Investigator (example. language problem, illiterates, poor mental status) or to comply with the requirements of the entire study, including dietary restrictions
* Vulnerable participants (example., persons kept in detention).
* Legal incapacity or limited legal capacity
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany, will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200585_0004
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 participants were randomized in 1:1 ratio to the two treatment sequences: Sequence 1 (First Cesol, Then Biltricide, Then Cesol and Then Biltricide) and Sequence 2 (First Biltricide, Then Cesol, Then Biltricide and Then Cesol).
Groups:
- First Cesol, Then Biltricide, Then Cesol and Then Biltricide: Participants received first single oral dose of 1200 milligrams (mg) (two 600 mg film-coated tablets) Cesol (Test 1) on Day 1 in treatment period 1 followed by first single oral dose of 1200 mg (two 600 mg film-coated tablets) Biltricide (Reference 1) on Day 8 in treatment period 2 followed by second single oral dose of 1200 mg (two 600 mg film-coated tablets) Cesol (Test 2) on Day 15 in treatment period 3 followed by second single oral dose of 1200 mg (two 600 mg film-coated tablets) Biltricide (Reference 2) on Day 22 in treatment period 4 under fed conditions. A washout period of 7 days was maintained between 4 treatment periods.
- First Biltricide, Then Cesol, Then Biltricide and Then Cesol: Participants received first single oral dose of 1200 mg (two 600 mg film-coated tablets) Biltricide (Reference 1) on Day 1 in treatment period 1 followed by first single oral dose of 1200 mg (two 600 mg film-coated tablets) Cesol (Test 1) on Day 8 in treatment period 2 followed by second single oral dose of 1200 mg (two 600 mg film-coated tablets) Biltricide (Reference 2) on Day 15 in treatment period 3 followed by second single oral dose of 1200 mg (two 600 mg film-coated tablets) Cesol (Test 2) on Day 22 in treatment period 4 under fed conditions. A washout period of 7 days was maintained between 4 treatment periods.
Period: Treatment Period 1
Arm/Group | First Cesol, Then Biltricide, Then Cesol and Then Biltricide | First Biltricide, Then Cesol, Then Biltricide and Then Cesol
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | First Cesol, Then Biltricide, Then Cesol and Then Biltricide | First Biltricide, Then Cesol, Then Biltricide and Then Cesol
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Treatment Period 3
Arm/Group | First Cesol, Then Biltricide, Then Cesol and Then Biltricide | First Biltricide, Then Cesol, Then Biltricide and Then Cesol
Started | 17 | 18
Completed | 16 | 17
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Treatment Period 4
Arm/Group | First Cesol, Then Biltricide, Then Cesol and Then Biltricide | First Biltricide, Then Cesol, Then Biltricide and Then Cesol
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | First Cesol, Then Biltricide, Then Cesol and Then Biltricide | First Biltricide, Then Cesol, Then Biltricide and Then Cesol | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (10.8) | 37 (10.8) | 34 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Racemic-Praziquantel (Rac-PZQ)
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 8.0, 9.0, 10.0 and 12 hours post-dose in each treatment period
Population: The Pharmacokinetic (PK) Analysis Set included all participants, who received at least one dose of study intervention, had no clinically important protocol deviations or important events affecting PK, and provided at least one measurable post-dose concentration. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Cesol First Administration: Participants who received single oral dose of 1200 mg (two 600 mg tablets) Cesol (Test 1) in either Treatment Period 1 or 2 under fed conditions.
- Cesol Second Administration: Participants who received single oral dose of 1200 mg (two 600 mg tablets) Cesol (Test 2) in either Treatment Period 3 or 4 under fed conditions.
- Biltricide First Administration: Participants who received single oral dose of 1200 mg (two 600 mg tablets) Biltricide (Reference 1) in either Treatment Period 1 or 2 under fed conditions.
- Biltricide Second Administration: Participants who received single oral dose of 1200 mg (two 600 mg tablets) Biltricide (Reference 2) in either Treatment Period 3 or 4 under fed conditions.
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
nanogram per milliliter (ng/mL) | 421 (118.3) | 415 (129.1) | 425 (98.3) | 459 (129.5)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Racemic-Praziquantel (Rac-PZQ)
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: as for outcome 1
Population: The PK Analysis Set included all participants, who received at least one dose of study intervention, had no clinically important protocol deviations or important events affecting PK, and provided at least one measurable post-dose concentration. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
hours*nanogram per milliliter (h*ng/mL) | 894 (114.6) | 873 (118.9) | 886 (105.7) | 964 (124.8)

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Related TEAEs
Description: Adverse event (AE): any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: AE with onset after start of treatment or with onset date before the treatment start date but worsening after the treatment start date. TEAEs included both serious and non-serious TEAEs. Treatment-related TEAEs: reasonably related to the study intervention. Number of participants with TEAEs and treatment related TEAEs were reported.
Time Frame: Baseline up to Day 27
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 36 | 34
Participants
  TEAEs | 6 | 6 | 7 | 7
  Treatment related TEAEs | 6 | 6 | 7 | 6

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) by Severity According to Qualitative Toxicity Scale
Description: Severity of TEAEs were graded using Qualitative Toxicity Scale, as follows: Mild: Participant is aware of the event or symptom, but the event or symptom is easily tolerated; Moderate: Participant experiences sufficient discomfort to interfere with or reduce his or her usual level of activity; Severe: Significant impairment of functioning: the participant is unable to carry out his or her usual activities. Number of participants with TEAEs by severity were reported.
Time Frame: Baseline up to Day 27
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 36 | 34
Participants
  Mild TEAEs | 5 | 5 | 5 | 5
  Moderate TEAEs | 2 | 1 | 4 | 2
  Severe TEAEs | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Relevant Changes From Baseline in Laboratory Parameters
Description: Laboratory investigation included hematology, biochemistry and urinalysis. Clinical relevance was determined by the investigator. The number of participants with clinically relevant changes from baseline in laboratory parameters were reported.
Time Frame: Baseline up to Day 27
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 36 | 34
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Relevant Changes From Baseline in Vital Signs
Description: Vital signs included body temperature, systolic and diastolic blood pressure and pulse rate. Clinical relevance was determined by the investigator. The number of participants with clinically relevant changes from baseline in vital signs were reported.
Time Frame: Baseline up to Day 27
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Biltricide Second Administration: Participants who received single oral dose of 1200 mg (two 600 mg tablets) Biltricide (Reference 2) in either Treatment Period 1 or 2 under fed conditions.
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 36 | 34
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Findings
Description: 12-lead ECG recordings included rhythm, heart rate (as measured by RR interval), PR interval, QRS duration and QT interval. The corrected QT interval (QTcF) was calculated using Fridericia's formula. 12-lead ECG recordings were obtained after the participants have rested for at least 10 minutes in semisupine position. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in 12-Lead ECG findings were reported.
Time Frame: Baseline up to Day 27
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 36 | 34
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Praziquantel (PZQ) Enantiomers: R-(-)-PZQ and S-(+) PZQ
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
ng/mL
  R-(-)-PZQ | 67.8 (148.3) | 71.4 (138.8) | 66.2 (132.9) | 80.0 (176.2)
  S-(+)-PZQ | 349 (114.3) | 346 (123.2) | 355 (94.4) | 374 (122.2)

9. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Praziquantel (PZQ) Enantiomers: R-(-)-PZQ and S-(+)-PZQ
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
h*ng/mL
  R-(-)-PZQ | 103 (204.9) | 111 (146.5) | 104 (153.9) | 125 (190.9)
  S-(+)-PZQ | 772 (110.9) | 758 (115.4) | 767 (104.3) | 824 (118.9)

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Racemic-Praziquantel (Rac-PZQ), R-(-)-PZQ and S-(+)-PZQ
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: as for outcome 1
Population: The PK Analysis Set included all participants, who received at least one dose of study intervention, had no clinically important protocol deviations or important events affecting PK, and provided at least one measurable post-dose concentration. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable for the specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
h*ng/mL
  rac-PZQ | 932 (113.4) | 907 (117.0) | 926 (104.7) | 1001 (123.8)
  R-(-)-PZQ: number analyzed (Participants) | 28 | 27 | 29 | 28
  R-(-)-PZQ | 175 (115.1) | 166 (97.9) | 157 (94.9) | 179 (145.7)
  S-(+)-PZQ | 813 (111.6) | 792 (114.0) | 808 (103.7) | 864 (118.7)

11. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Racemic-Praziquantel (Rac-PZQ), R-(-)-PZQ and S-(+)-PZQ
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
hours
  rac-PZQ | 2.50 [0.500 to 3.50] | 2.00 [0.500 to 4.00] | 2.50 [0.500 to 5.00] | 2.50 [0.500 to 4.50]
  R-(-)-PZQ: number analyzed (Participants) | 36 | 33 | 35 | 34
  R-(-)-PZQ | 2.50 [0.500 to 3.50] | 2.00 [0.500 to 3.50] | 2.50 [0.500 to 5.00] | 2.50 [0.250 to 4.50]
  S-(+)-PZQ | 2.50 [0.500 to 3.50] | 2.00 [0.500 to 4.00] | 2.50 [0.500 to 5.00] | 2.50 [0.500 to 4.50]

12. Secondary Outcome: Time Prior to the First Measurable (Non-zero) Concentration (Tlag) of Racemic-Praziquantel (Rac-PZQ), R-(-)-PZQ and S-(+)-PZQ
Description: Time prior to the first measurable (non-zero) concentration; calculated as last time point at which the concentration is less than (<) Lower Limit of Quantification (LLQ) before the occurrence of the first quantifiable concentration.
Time Frame: as for outcome 1
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
hours
  rac-PZQ | 0.750 [0.00 to 2.50] | 0.500 [0.00 to 2.50] | 1.00 [0.00 to 2.00] | 0.750 [0.00 to 2.50]
  R-(-)-PZQ: number analyzed (Participants) | 36 | 33 | 35 | 34
  R-(-)-PZQ | 1.00 [0.00 to 3.00] | 1.00 [0.00 to 3.00] | 1.00 [0.00 to 2.50] | 1.00 [0.00 to 2.57]
  S-(+)-PZQ | 0.750 [0.00 to 2.50] | 0.500 [0.00 to 2.50] | 1.00 [0.00 to 2.00] | 0.750 [0.00 to 2.50]

13. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of Racemic-Praziquantel (Rac-PZQ), R-(-)-PZQ and S-(+)-PZQ
Description: Elimination Half Life (T1/2) was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. T1/2 was calculated by natural log 2 divided by Lambda z. Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: as for outcome 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
hours
  rac-PZQ | 2.44 (4.00) | 2.08 (47.3) | 2.43 (47.9) | 2.20 (49.4)
  R-(-)-PZQ: number analyzed (Participants) | 28 | 27 | 29 | 28
  R-(-)-PZQ | 1.39 (61.5) | 1.35 (48.8) | 1.35 (53.7) | 1.24 (54.4)
  S-(+)-PZQ | 2.62 (43.6) | 2.18 (48.5) | 2.51 (47.2) | 2.34 (51.7)

14. Secondary Outcome: Terminal Rate Constant (Lambda z) of Racemic-Praziquantel (Rac-PZQ), R-(-)-PZQ and S-(+)-PZQ
Description: Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: as for outcome 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
1/hour
  rac-PZQ | 0.284 (40.0) | 0.334 (47.3) | 0.285 (47.9) | 0.315 (49.4)
  R-(-)-PZQ: number analyzed (Participants) | 28 | 27 | 29 | 28
  R-(-)-PZQ | 0.499 (61.5) | 0.514 (48.8) | 0.515 (53.7) | 0.559 (54.4)
  S-(+)-PZQ | 0.265 (43.6) | 0.318 (48.5) | 0.276 (47.2) | 0.297 (51.7)

15. Secondary Outcome: Apparent Clearance (CL/f) of Racemic-Praziquantel (Rac-PZQ), R-(-)-PZQ and S-(+)-PZQ
Description: CL/f was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. CL/f was calculated as Dose/AUC0-inf, where AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. AUC0-inf was calculated as AUC0-t + Clast pred/Lambda Z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the lower limit of quantification (LLQ) and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
liter per hour
  rac-PZQ | 1287 (113.4) | 1323 (117.0) | 1296 (104.7) | 1199 (123.8)
  R-(-)-PZQ: number analyzed (Participants) | 28 | 27 | 29 | 28
  R-(-)-PZQ | 6868 (115.1) | 7251 (97.9) | 7620 (94.9) | 6700 (145.7)
  S-(+)-PZQ | 1475 (111.6) | 1516 (114.0) | 1486 (103.7) | 1389 (118.7)

16. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/f) of Racemic-Praziquantel (Rac-PZQ), R-(-)-PZQ and S-(+)-PZQ
Description: Vz/f: the distribution of a study drug between plasma and the rest of the body after oral dosing. For single dose Vz/f = Dose/(AUC0-inf*Lambda Z), where AUC0-inf = (AUC0-t + Clast pred/Lambda Z). Clastpred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and Lambda Z = the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 36 | 34 | 35 | 34
liters
  rac-PZQ | 4528 (99.9) | 3963 (87.5) | 4542 (98.6) | 3801 (110.5)
  R-(-)-PZQ: number analyzed (Participants) | 28 | 27 | 29 | 28
  R-(-)-PZQ | 13761 (70.3) | 14100 (63.4) | 14806 (56.8) | 11993 (83.7)
  S-(+)-PZQ | 5568 (79.6) | 4765 (82.0) | 5385 (89.1) | 4685 (97.1)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 27
Description: The Safety Analysis Set included all participants who were administered any dose of any study intervention.
Arm/Group | Cesol First Administration | Cesol Second Administration | Biltricide First Administration | Biltricide Second Administration
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34 | 0/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34 | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 6/36 | 6/34 | 7/36 | 7/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cesol First Administration (N=36) | Cesol Second Administration (N=34) | Biltricide First Administration (N=36) | Biltricide Second Administration (N=34)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 6 | 5
Body temperature increased (Investigations) | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT04314037/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT04314037/SAP_001.pdf